CLINICAL TRIAL: NCT03023865
Title: Individualized Diagnosis and Treatment for Long Gap Esophageal Atresia Based on the Principle of Biological Growth Under Stress
Brief Title: Individualized Management for Long Gap Esophageal Atresia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XH-16-033
Record Dates: First submitted 2016-10-26; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-10

CONDITIONS: Esophageal Atresia
Keywords: Long gap esophageal atresia
MeSH Terms: conditions — Esophageal Atresia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Staged stress function (Experimental): A preoperative staged stress function procedure for elongation of the proximal and distal segments to achieve utilizing the native esophagus to establish esophageal continuity
  Interventions: Procedure: Staged stress function

INTERVENTIONS:
Procedure: Staged stress function — A preoperative staged stress function procedure for elongation of the proximal and distal segments to achieve utilizing the native esophagus to establish esophageal continuity

SUMMARY:
The treatment of long gap esophageal atresia (LGEA) in neonates is one of the most challenging congenital malformations in neonatal surgery. Usually the proximal and distal segments of the esophagus are too far apart, which leads to primary anastomosis abandoned. Thus various techniques have been used including Circular and spiral myotomies、Foker and Kimura elongation and gastrointestinal replacement. They are being widely used but bring more complications and less effectiveness. And considering about the absence of definite guideline for the diagnosis and treatment of LGEA worldwide, We prepare to use a preoperative staged stress function procedure for elongation of the proximal and distal segments, then to obtain an exact evaluation of the pouch status to achieve an individualized protocol of diagnosis and treatment utilizing the native esophagus to establish esophageal continuity for patients with LGEA.

DETAILED DESCRIPTION:
Patients with diagnosis of LGEA(gap distance>3.5cm) will be accepted to the program.

After accepted to our center, the patients will feed by gastrostomy tube to keep nutritional status remain well controlled. Continuous suction in the upper pouch will be applied to avoid aspiration pneumonia.

We will design a bouginage with baroreceptor. Then the stress function will be performed as following steps. The designed bouginage will be inserted into the upper esophagus pouch through oral cavity with a certain downward longitudinal force to increase esophageal length by tissue stretch and growth, it will be performed 10-15 minutes each time once/twice a day. While the elongation of distal pouch will be achieved via the gastrostomy using the same bouginage to give upward pressure, the program will be operated under X-ray firstly to avoid injury or false passage formation,it can be performed in the ward thereafter. The gap length and the diameter of the pouch will be evaluated every 1-2 weeks. During the elongation period, continuous upper pouch suctioning and nutritional support were maintained.

When the gap distance is short enough，the method of surgery will be decided，including end-to-end anastomosis、Livadites、flip-flap and choice of thoracoscopy use. The purpose of the program is to achieve the exact management and treatment for patients with LGEA and help promoting the use of the new technology.

ELIGIBILITY:
Inclusion Criteria：

* Patients with long gap esophageal atresia（LGEA）which the gap lenth≥3.5cm；
* with（out）tracheoesophageal fistula（TEF）

Exclusion Criteria:

* Patients with LGEA which can not accept the staged stress function

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with LGEA cured by the elongation method | up to 3 years
  Provide the numbers of patients with LGEA cured by the method using elongation technique

SECONDARY OUTCOMES:
Data collection of patients with LGEA | up to 3 years
  Circumstances of diagnosis，gap length in centimetre between esophageal pouches ，operation method，modalities in percent of follow-up clinical management

CONTACTS AND LOCATIONS:
Overall Officials: Wang Jun, MD, Study Director — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Department of Pediatric Surgery, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Share with the period of stress applied,gap distance between two esophageal segments,stress pressure.etc

REFERENCES:
- [Background] von Allmen D, Wijnen RM. Bridging the Gap in the Repair of Long-Gap Esophageal Atresia: Still Questions on Diagnostics and Treatment. Eur J Pediatr Surg. 2015 Aug;25(4):312-7. doi: 10.1055/s-0035-1562926. Epub 2015 Aug 24. PMID 26302063
- [Background] Spitz L, Kiely EM, Drake DP, Pierro A. Long-gap oesophageal atresia. Pediatr Surg Int. 1996 Aug;11(7):462-5. doi: 10.1007/BF00180083. Epub 2013 Sep 21. PMID 24057783
- [Background] Rothenberg SS, Flake AW. Experience with Thoracoscopic Repair of Long Gap Esophageal Atresia in Neonates. J Laparoendosc Adv Surg Tech A. 2015 Nov;25(11):932-5. doi: 10.1089/lap.2015.0124. Epub 2015 Oct 20. PMID 26485521